CLINICAL TRIAL: NCT05416112
Title: Non Invasive Left Ventricle Contractility dp/dt Could be Used as a Prognostic Marker in Patients Admitted to the Emergency Department for Chest Pain
Brief Title: Non-invasive Left Ventricle Contractility dp/dt as Prognostic Marker in Chest Unit Patients
Acronym: dp/dt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Other Study IDs: dp/dt
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chest Pain
Keywords: chest pain,; myocardial ischemia,; acute myocardial dysfunction,; plethysmography,; non invasive dp/dt.
MeSH Terms: conditions — Chest Pain; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ischemic heart disease is a major public health problem with high mortality rate despite the progress in management and the resources mobilized. The idea is that myocardial ischemia is generally associated with left ventricular dysfunction and, consequently, a possible alteration of the dp/dt index. As dp/dt could be assessed non-invasively by plethysmographic method, it is interesting to investigate its prognostic performance in patients with indifferentiate chest pain.

DETAILED DESCRIPTION:
Ischemic heart disease remains a major public health problem. Despite all the advances in the prognostic approach to ischemic heart disease, the risk of occurrence of major cardiovascular events is not negligible. Several scores have been proposed for chest pain stratification risk, the most widely used are the TIMI and the GRACE scores.

The dP/dt max is therefore an excellent index of contractility, corresponding to the maximum level of tension developed by an isolated cardiac muscle during the isovolumic contraction phase.

the investigator theorized that a less value of dp/dt would be associated with more major cardiovascular events (MACE), because ischemia reduces myocardial contractility.

The current study describes non-invasive plethysmographic dp/dt changes, which could be used as a prognostic marker in patients presenting at the emergency department with acute chest pain.

ELIGIBILITY:
Inclusion criteria:

* age over 18 years old,
* acute chest pain

Exclusion criteria:

* traumatic chest pain,
* hemodynamic instability;
* arrhythmias;
* holders of a pacemaker;
* STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting to the emergency department with acute chest pain
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
MACE | one month
  the occurrence of a major cardiovascular event (MACE)
MACE | SIX MONTHS
  : the occurrence of a major cardiovascular event (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, professor, Principal Investigator — Monastir University Hospital, Monastir, Tunisia, 5000
Locations (1):
- Emergency Departement, Monastir, Tunisia